CLINICAL TRIAL: NCT03513627
Title: Comparison of Microvascular Reactivity Assessed by Post-occlusive Reactive Hyperaemia Test in Gingiva at Natural Tooth and at Implant Borne Crown
Brief Title: Microvascular Reactivity of the Gingiva Around Implant Born Crown
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: 4/2018
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Dental Implants
Keywords: periimplant soft tissue; gingiva; human; microcirculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Implant: Post-occlusive reactive hyperaemia test (PORH test) in the gingiva at a dental implant born crown in the front region of the jaw
  Interventions: Procedure: Post-occlusive reactive hyperemia test (PORH test)
- Tooth: Post-occlusive reactive hyperaemia test (PORH test) in the gingiva at the contralateral natural tooth
  Interventions: Procedure: Post-occlusive reactive hyperemia test (PORH test)

INTERVENTIONS:
Procedure: Post-occlusive reactive hyperemia test (PORH test) — Compression is applied on the buccal side of the attached gingiva, perpendicular to the long axis of the natural or implant born crown 2 mm far from the gingival margin.

SUMMARY:
Apply LSCI method for follow-up changes in regional blood flow after compression of the gingiva in order to compare the vascular reactivity of the attached gingiva at implant versus at tooth.

DETAILED DESCRIPTION:
This study will examine the effects of implantation and peri-implant soft tissue shaping on the circulation and the regeneration processes of the human gingiva.

The primary aim is to determine the effect of a short term disruption of the blood flow in the gingiva next to an implant and the contralateral tooth, in order to compare the functionally active collateral circulation in the attached gingiva at these respective regions. Using Laser Speckle Contrast Imaging technique (LSCI), which provides blood perfusion data, the investigators will have the possibility to detect functional alterations in gingival microcirculation during and after a short term compression of the gingiva. The secondary aim is to assess and compare the time course of the restoration of the circulation on the affected areas. Further aims are to observe if the compensation capability of the circulation is influenced by gingival thickness (biotype) and patient's gender.

ELIGIBILITY:
Inclusion Criteria:

Patient with single dental implant installed in the front region of the jaw at least 6 months ago. On the contralateral side a natural tooth is located.

Exclusion Criteria:

* systemic disease
* smoking
* alcohol abuse
* pregnancy
* gingivitis
* periodontitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy patients who are not taking medication, with healthy gingiva
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Magnitude of the hyperemia after PORH test | 5min
  Blood flow changes are measured by LSCI before (baseline), during and after gingiva compression. The scale is an arbitrary unit (0-3000 LSPU); relative changes to the baseline measurement will be calculate.

SECONDARY OUTCOMES:
Longevity of the hyperemia after PORH test | 20min
  Blood flow changes are measured by LSCI before (baseline), during and after gingiva compression. The scale is an arbitrary unit (0-3000 LSPU); relative changes to the baseline measurement will be calculate.
Size of the hyperemia after PORH test | 20 min
  Blood flow changes are measured by LSCI before (baseline), during and after gingiva compression. LSCI can measure in several cm2 areas and display blood perfusion as color-coded images.
Difference in the magnitude and longevity of hyperemia induced by PORH test next to an implant born crown between women and men. | 20 min
  Blood flow changes are measured by LSCI before (baseline), during and after gingiva compression. The scale is an arbitrary unit (0-3000 LSPU); relative changes to the baseline measurement will be calculate.

CONTACTS AND LOCATIONS:
Locations (1):
- Janos Vag, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No